CLINICAL TRIAL: NCT05432492
Title: A Phase II Study of AK112 (PD-1/VEGF Bispecific) in Patients With Unresectable Hepatocellular Carcinoma (HCC)
Brief Title: A Study of AK112 in Patients With Unresectable Hepatocellular Carcinoma (HCC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK112-207
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Subjects receive AK112 on Day 1 of every 3-week cycle (Q3W) until progression.
  Interventions: Drug: AK112
- Cohort 2 (Experimental): Subjects receive AK112 on Day 1 of every 3-week cycle (Q3W) until progression.
  Interventions: Drug: AK112

INTERVENTIONS:
Drug: AK112 — IV infusion, specified dose on specified days

SUMMARY:
Phase II open label, multicenter study to evaluate the efficacy and safety of AK112 (PD-1/VEGF Bispecific) in patients with unresectable hepatocellular carcinoma (HCC).

ELIGIBILITY:
Inclusion Criteria:

* Be able and willing to provide written informed consent and to comply with all requirements of study participation (including all study procedures).
* 18 to 75 years old.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Have a life expectancy of at least 3 months.
* BCLC stage B or C, not amenable to curative surgery.
* Hepatocellular carcinoma confirmed by histology/cytology. Cirrhosis meets the clinical diagnostic criteria for hepatocellular carcinoma of the American Association for the Diagnosis of Liver Diseases (AASLD).
* At least one measurable untreated lesion.
* Child-Pugh class A.
* Has adequate organ function.
* All female and male subjects of reproductive potential must agree to use an effective method of contraception, as determined by the Investigator, during and for 120 days after the last dose of study treatment.

Exclusion Criteria:

* With fibrous lamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, cholangiocarcinoma components in tumor tissues.
* History of malignancy other than HCC within 5 years, except that basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Have a history of hepatic encephalopathy or have a history of liver transplantation.
* With clinical symptoms requires drainage of pleural effusion, ascites or pericardial effusion.
* Central nervous system (CNS) metastasis or meningeal metastasis.
* Prior immunotherapy with an anti-PD-1, anti-PD-L1, or anti-CTLA-4 antibody (or any other antibody or drug specifically targeting T-cell costimulation or checkpoint pathways).
* Prior systemic bevacizumab and its analogues treatment.
* Severe bleeding tendency or coagulation dysfunction; occurred arteriovenous thromboembolic events or bleeding events due to esophageal and/or gastric varices within 6 months before the first administration.
* Known presence or history of required hormone treatment interstitial lung disease or non-infectious pneumonitis.
* Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has undergone major surgery within 30 days prior to the first dose of study treatment.
* History of myocardial infarction, unstable angina, cardiac or other vascular stenting, angioplasty, or surgery within 12 months.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Number of patients with Adverse Events (AEs) | Up to approximately 2 years
Objective Response Rate (ORR) Per RECIST v1.1 | Up to approximately 2 years
Objective Response Rate (ORR) Per mRECIST | Up to approximately 2 years

SECONDARY OUTCOMES:
Disease control rate (DCR) | Up to approximately 2 years
Duration of Response (DoR) | Up to approximately 2 years
Time to response (TTR) | Up to approximately 2 years
Progression free survival (PFS) | Up to approximately 2 years
Overall survival (OS) | Up to approximately 2 years

OTHER OUTCOMES:
Percentage of participants who obtain R0 resection | Up to approximately 2 years
Percentage of participants who obtain a major pathologic responses (MPR) | Up to approximately 2 years
Percentage of participants who obtain a pathologic complete response (pCR) | Up to approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jingfeng Liu, Principal Investigator — Fujian Cancer Hospital